CLINICAL TRIAL: NCT01521442
Title: Mindful Yoga Therapy as an Adjunctive Treatment for PTSD Among OEF/OIF Veterans: A Pilot Study
Brief Title: Mindful Yoga Therapy as an Adjunctive Treatment for PTSD Among OEF/OIF Veterans
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Did not have funding or resources to carry out study
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01540
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: PTSD
Keywords: PTSD; Yoga; Complementary and Alternative Medicine (CAM)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 12 sessions of Mindful Yoga Therapy delivered two times per week for 75 minutes each.
  Interventions: Behavioral: Mindful Yoga Therapy
- Arm 2 (Other): 12-week delay before beginning Mindful Yoga Therapy treatment which will consist of 12 sessions of Mindful Yoga Therapy delivered two times per week for 75 minutes each.
  Interventions: Behavioral: Wait-list Control

INTERVENTIONS:
Behavioral: Mindful Yoga Therapy — Veterans will participate in twice weekly Mindful Yoga Therapy, which includes meditation, breathing practices, mindful movement, and guided rest (yoga nidra), as well as daily home practice.
  Arms: Arm 1
Behavioral: Wait-list Control — Participants will receive Mindful Yoga Therapy intervention after 12 weeks from being enrolled. Veterans will participate in twice weekly Mindful Yoga Therapy, which includes meditation, breathing practices, mindful movement, and guided rest (yoga nidra), as well as daily home practice.
  Arms: Arm 2

SUMMARY:
The primary objective of the current study is to establish the safety and acceptability of Mindful Yoga Therapy as an adjunctive treatment for posttraumatic stress disorder (PTSD) among Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn (OEF/OIF/OND) Veterans. The current study also seeks to establish preliminary efficacy of Mindful Yoga Therapy for reduction of symptoms of PTSD and explore heart rate variability as a mechanism of therapeutic action.

DETAILED DESCRIPTION:
PTSD is a chronic, debilitating anxiety disorder associated with disability, functional impairment, and a host of co-morbid physical and mental health conditions. Although several treatments are successful in treating Veterans with PTSD, many Veterans fail to complete these treatments and many others complete treatment without significant relief from symptoms. Yoga is one integrative treatment option that has shown promise for a number of physical and mental health conditions, including the treatment of depressive and anxiety disorders in civilian samples, and chronic pain in Veterans. Yoga is widely offered in Veterans Affairs (VA) PTSD Treatment Programs, yet there is a lack of research on its efficacy for PTSD in Veterans.

Mindful Yoga Therapy (MYT)is a 12-week treatment protocol incorporating meditation, breathing exercises, mindful movement practice, and guided rest (yoga nidra) that has been developed specifically for Veterans with PTSD. This pilot randomized clinical trial with cross-over waitlist comparison (RCT) will compare Immediate Mindful Yoga Therapy (MYT) plus Treatment as Usual (TAU) with Delayed MYT + TAU. Baseline (week 0), 12-week, and 24-week assessments, in addition to 36-week assessments for the delayed MYT treatment group, will include diagnostic, neurocognitive, and psychophysiological measures conducted by a research team member blinded to treatment condition.

Primary Aim: The primary aim of the current pilot study is to establish the safety and acceptability of Mindful Yoga Therapy as an adjunctive treatment for PTSD among OEF/OIF Veterans.

Specific Aim #1: To establish that MYT is a treatment that can be implemented safely. Hypothesis #1: There will be no significant difference in the number of adverse events between treatment groups from week 0 to week 12.

Specific Aim #2: To establish that MYT is a treatment that veterans find helpful and accessible. Hypothesis #2. At least 50% of participants completing the MYT treatment will report that the treatment was helpful and accessible as reported on self-report measures of treatment satisfaction, administered at the completion of the MYT treatment component of the study (week 12 for the immediate MYT treatment group; week 24 for the delayed MYT treatment group).

Secondary Aim: To assess the effect of Mindful Yoga Therapy as an adjunctive treatment on symptoms of PTSD is OEF/OIF Veterans.

Specific Aim #3: To examine the efficacy of MYT + TAU in reducing frequency and/or intensity of PTSD symptoms. Hypothesis #3. While both groups are expected to show reductions in symptoms, compared to participants in the Delayed MYT + TAU group, Veterans in the Immediate MYT + TAU group will exhibit significantly greater reductions in the frequency and/or intensity of PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS) (baseline to 12-week change). We predict that Immediate MYT+TAU will have a differential impact on the three PTSD symptom clusters, with the greatest effect on the hyperarousal symptoms.

Specific Aim #4. To document the durability of MYT treatment effects in the Immediate MYT group. Hypothesis #4. PTSD symptom scores will not be significantly different at 24-week assessment compared to those at week 12 assessment in the immediate MYT treatment group, and not significantly different at 36-week assessment compared to 24-week assessment for the delayed treatment group.

Tertiary Aim: To assess changes in heart rate variability from a resting baseline period and a guided meditation period in Veterans with PTSD before and after treatment with Mindful Yoga Therapy.

Specific Aim #5: To examine the predictive value of HRV on outcomes of Immediate MYT+TAU and Delayed MYT + TAU. Hypothesis #5. Increases in high frequency HRV (HF-HRV) from resting baseline to guided meditation at the pre-treatment assessment (week 0 for the immediate MYT treatment group, week 12 for the delayed MYT treatment group) will be associated with greater PTSD symptom reduction at post-treatment (week 12 for the immediate MYT treatment group; week 24 for delayed MYT treatment group).

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veteran
* Ages 18-45
* Currently enrolled in active PTSD treatment
* Meet criteria for PTSD
* Veteran with combat exposure during deployment

Exclusion Criteria:

* Current psychotic disorder or bipolar disorder
* Current use of beta-blocker medication
* Current regular yoga or meditation practice in the past month
* Significant limitations or injuries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | 12 weeks
  The "gold standard" measure of frequency and intensity of PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Heapy, Ph.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States